CLINICAL TRIAL: NCT04928573
Title: Retrospective Observational Study for Late Assessment of the Safety and Efficacy of Biosimilar Rituximab: a Subanalysis of the RTXM83-AC-01-11 Trial
Brief Title: Study for Late Assessment of the Safety and Efficacy of Biosimilar Rituximab
Status: Completed | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB2002
Record Dates: First submitted 2021-05-28; First posted 2021-06-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: rituximab; Vivaxxia; Diffuse Large B Cell Lymphoma; biosimilar
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I: All participants previously randomized in Brazil for the phase III study RTXM83-AC-01-11 already completed, which was conducted to support the registration of the new biosimilar of rituximab (Vivaxxia) in different countries.
  The RTXM83-AC-01-11 study compared the efficacy and safety between biosimilar rituximab (RTXM83) and the reference rituximab (Mabthera®), both associated with CHOP chemotherapy (RTXM83-CHOP and R-CHOP, respectively) and included participants of the research with a diagnosis of lymphoma other than large B cell (LDGCB) CD20 positive.

SUMMARY:
The RTXM83-AC-01-11 study evaluated efficacy and safety outcomes in relation to the use of Vivaxxia during 6 treatment cycles (at the investigator's discretion, up to 8 treatment cycles could be administered), followed by 9 months of follow-up. , this follow-up time being sufficient for the analysis of non-inferiority in relation to the reference medicine. However, data on late events of efficacy and safety are of great value to contribute to a robust clinical response and to strengthen confidence in the use of biosimilar medicines. For this reason, Libbs Farmacêutica proposes this retrospective observational study to collect data on late outcomes of the pivotal study that directed the approval of the biosimilar rituximab (Vivaxxia) from the research participants from Brazil.

The present retrospective observational study LB2002 will sub-analyze selected results of efficacy and safety from study RTXM83-AC-01-11 in participants over 18 years of age randomized in Brazil, totaling 28 participants, in addition to evaluating late efficacy and safety outcomes. Information on subsequent treatment / protocol should also be collected for participants who have progressive or recurrent disease, instituted by research centers under these conditions.

The proposal is to compare descriptively the selected outcomes of efficacy and safety of these participants with the same outcomes selected for the global population in the RTXM83-AC-01-11 study, and also provide late safety and effective data important for anti-neoplastic processes.

DETAILED DESCRIPTION:
Evaluate research participants who were refractory to treatment, defined as not having achieved: Complete Response (CR) or Partial Response (PR), after 6 treatment cycles in study RTXM83-AC-01-11.

Evaluate the participants who had a recurrence of the disease, defined as a change from: Complete Response (CR), after 06 treatment cycles in study RTXM83-AC-01-11, to: Progressive Disease (PD) until the date of consent (ICF) in the LB2002 study.

The data of the subsequent treatment / protocol instituted by the research center for progressive or recurrent disease will also be collected.

PERIOD OF ANALYSIS OF THIS CLINICAL STUDY

* 01-JUL-2013 (beginning of the study) to 17-JUL-2017 (data in which the last participant of the study RTXM83-AC-01-11 arrived at the last follow-up visit at 9 months after the last dose of treatment): for sub-analysis of efficacy and safety proposed by study RTXM83-AC-01-11: SLE, TRG and EA, and for exploratory evaluation of refractory disease.
* Data from randomization in study RTXM83-AC-01-11 to consent data (TCLE) in study LB2002: for analysis of SLP, SG and for exploratory evaluation of relapse.
* Date of the final visit of study RTXM83-AC-01-11, considered as FUP3, until the date of consent (ICF) in study LB2002: for the evaluation of late AEs of interest.

Data collect:For the subanalysis evaluations, the data that have already been collected will be used and are part of the study database RTXM83-AC-01-11. This database will also be considered for exploratory assessment of refractory disease.

For late evaluations of safety and efficacy (late adverse events of interest, SLP, SG and disease recurrence) and also data on the subsequent treatment / protocol instituted by the research center for progressive disease or disease recurrence, data from medical records available at research centers.

Finally, all the data necessary to evaluate the objectives established in this study will be imputed in a single Electronic Case Report Form (eCRF) developed exclusively for this project.

ELIGIBILITY:
Inclusion Criteria:

* Free and informed consent to participate in this retrospective, observational study of data collection
* Research participants from Brazil randomized and who received at least one dose of treatment in the RTXM83-AC-01-11 study.

Exclusion Criteria:

* not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants previously randomized in Brazil for the phase III study RTXM83-AC-01-11, already completed, will be eligible for this observational, retrospective study LB2002, which was conducted to support the registration of the new biosimilar of rituximab (Vivaxxia) in different countries.
  The RTXM83-AC-01-11 study compared the efficacy and safety between biosimilar rituximab (RTXM83) and reference rituximab (Mabthera®), both associated with CHOP chemotherapy (RTXM83-CHOP and R-CHOP, respectively) and included participants of the research with a diagnosis of diffuse large B cell lymphoma (LDGCB) CD20 positive.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Effectiveness evaluation: subanalysis of event-free survival | 9 months after treatment
  To present the subanalysis of event-free survival of participants from Brazil in the two treatment groups (RTXM83-CHOP and R-CHOP) from the randomization date until the final visit of the RTXM83-AC-01-11 study, considered as o FUP 3 (9-month follow-up after the end of treatment);
Effectiveness evaluation: subanalysis of the Global Response Rate | At the end of Cycle 6 (each cycle is 03 weeks)
  To present the subanalysis of the Global Response Rate of participants from Brazil in the two treatment groups (RTXM83-CHOP and R-CHOP), after 6 treatment cycles in the RTXM83-AC-01-11 study, assessed as Complete Response ( RC) or Partial Response (PR);
Security evaluation: sub-analysis of the adverse events | 9 months after treatment
  Present the sub-analysis of the adverse events (AE) of the participants in Brazil that occurred from the date of signing the Free and Informed Consent Form (ICF) until the final visit of the study RTXM83-AC-01-11, considered as the FUP 3 (follow-up) 9 months after the end of treatment);
Effectiveness evaluation: progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months
  Assess progression-free survival in the two treatment groups (RTXM83-CHOP and R-CHOP) from the date of randomization in the RTXM83-AC-01-11 study until the date of consent (ICF) in the LB2002 study;
Effectiveness evaluation: Assess the overall survival | From date of randomization until the date of death from any cause, assessed up to 96 months
  Assess the overall survival in the two treatment groups (RTXM83-CHOP and R-CHOP) from the date of randomization in study RTXM83-AC-01-11 until the date of consent (ICF) in study LB2002;
Security evaluation: occurrence of late adverse events | From date of randomization until the date of death from any cause, assessed up to 96 months
  Evaluate the occurrence of late adverse events of interest from the date of the final visit of the RTXM83-AC-01-11 study, considered as FUP 3, until the date of consent (TCLE) in the LB2002 study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Fernando Pericole, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Delamain MT, Cardoso ACF, Pericole FV, da Silva Araujo SS, Fogliatto L, Higashi M, Pereira J, da Silva RL, Werutsky G, de Paulo Giacon Radtke P, Salvino MA, Castilho V. Long-Term Safety and Effectiveness of Rituximab Biosimilar RTXM83: A Retrospective Extension Study in Brazilian Patients with Diffuse Large B-Cell Lymphoma. Oncol Ther. 2024 Sep;12(3):585-598. doi: 10.1007/s40487-024-00282-7. Epub 2024 Jun 3. PMID 38829416